CLINICAL TRIAL: NCT02016326
Title: A Randomized Controlled Trial Comparing High-definition White Light Colonoscopy to I-scan Enhanced Colonoscopy for Adenoma Detection in a Population at Increased Risk of Colorectal Cancer (Main Study)
Brief Title: I-Scan Vs High Definition White Light (Main Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Robert Hilsden, Associate Professor, Department of Medicine & Research Director, Colon Cancer Screening Centre, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23474-M
Record Dates: First submitted 2013-11-13; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer
Keywords: Colonoscopy; High Definition White Light; I-Scan; Adenomas
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HD Colon (Experimental): High Definition White Light modality will be used by the endoscopist for the entire procedure.
  Interventions: Device: HD Colon
- I-Scan 1 (Experimental): I-scan 1 modality will be used by the endoscopist for the entire procedure.
  Interventions: Device: I-scan 1
- I-Scan 2 (Experimental): I-Scan 2 modality will be used by the endoscopist through out the procedure.
  Interventions: Device: I-Scan 2

INTERVENTIONS:
Device: HD Colon — High Definition White Light
  Arms: HD Colon
Device: I-scan 1 — I-Scan 1 has Contrast Enhancement(CE), Surface Enhancement(SE). SE mode highlights light-dark contrast thereby providing more mucosal surface detail. CE mode digitally adds blue to darker areas providing detailed imaging of subtle mucosal irregularities.
  Arms: I-Scan 1
Device: I-Scan 2 — I-Scan 1 has Contrast Enhancement(CE), Surface Enhancement(SE)and Tone Enhancement(TE). SE mode highlights light-dark contrast thereby providing more mucosal surface detail. CE mode digitally adds blue to darker areas providing detailed imaging of subtle mucosal irregularities. TE provides a uniform color image and is intended for detailed inspection of distinct lesions.
  Arms: I-Scan 2

SUMMARY:
The purpose of this study is to assess whether the use of I-Scan during colonoscopy leads to an increased yield of adenomas in the colon among a population at increased risk for CRC.

Primary Outcome:

Adenoma Detection Rate (ADR - No. of colonoscopies at which one or more histologically confirmed adenomas were found divided by the total no. of colonoscopies performed in the same time period) in the right colon using High Definition White Light Colonoscopy Versus I-Scan enhanced Colonoscopy.

Secondary Outcomes:

* Adenoma Detection Rate (ADR) of High Definition White Light Colonoscopy Versus I-Scan colonoscopy through out the entire colon.
* Adenoma Detection Rate (ADR) in the right colon during the "Second look", irrespective of imaging modality.
* Polyp Detection Rate (PDR - No. of colonoscopies at which one or more polyps were found(regardless of the histological type) divided by the total no. of colonoscopies performed in the Same time period) for each arm of the study in Right colon and throughout the entire colon.
* Mean number of adenomas per procedure for each arm of the study in right colon and throughout the entire colon.
* Mean number of polyps per procedure for each arm of the study in right colon and throughout the entire colon.
* Number of neoplastic lesions for each arm of the study in the right colon and throughout the entire colon and number of neoplastic lesions missed on 1st pass of right colon.
* Proportion of patients with diminutive lesions (< 5 mm) in each arm of the study
* Proportion of patients with Flat lesions (height < 1/2 diameter) in each arm of the study
* Proportion of patients with Sessile Serrated Adenoma in each arm of the study
* Proportion of patients with invasive cancer in each arm of the study
* Presence or absence of learning effect while using this technology given that use of I-Scan may train the human eye to better identify adenomas even without image enhancement.

DETAILED DESCRIPTION:
Colorectal Cancer is the third most common cause of cancer in Canada with an estimated lifetime risk of developing the disease of 6-7%. Each year there are approximately 21,000 new cases and 9,100 deaths attributable to this disease. Colonoscopy is one of several methods recommended for Colorectal Cancer (CRC) screening by current guidelines. While colonoscopy is the most invasive, it offers high diagnostic accuracy and ability for therapy (biopsy and removal of adenomas) compared to other modalities. The emerging evidence regarding missed neoplastic lesions with colonoscopy has resulted in quality initiatives designed to improve colonoscopy performance. I-Scan (Pentax, Montvale, NJ) is a new method that uses post processing computer algorithms to revise the standard white light to highlight pit patterns and vascular surface patterns.The relevant I-scan settings in the colon are I-scan 1 and I-scan 2. The primary objective of the study is to compare the adenoma detection rate in the right colon using High-definition white light colonoscopy versus I-scan enhanced colonoscopy.

All patients referred for a screening colonoscopy at Forzani and MacPhail Colon Cancer Centre will be considered for enrollment.All eligible patients that are not part of another research study will be approached for enrollment into the study. During the pre-assessment at the clinic a study assistant will contact all the eligible patients to describe the study and provide an "Invitation to participate in a Research study" form. The study assistant will obtain a final consent if they agree. Those not interested will simply receive the Centre's standard protocol. There will be no coercion of any sort. Following Informed Consent, treatment allocation through computer generated randomization will be revealed. Patients will be allocated to one of the three study arms (HD Colon, I-scan 1 and I-Scan 2). Patients will receive a standard bowel preparation: Split dose Polyethylene Glycol (PEG) (2L at noon + 2L at 8 PM the day before) for morning procedures or (2L at 8Pm the day before and 2L at five hours before the procedure on the day of colonoscopy) for afternoon procedure. certified gastroenterologists will perform all of the procedures with the assistance of a nurse. The planned "second look" of the right colon will involve withdrawing from the Cecum to Hepatic flexure, then re-inserting to Cecum and finally withdrawing through the entire colon. The physician performing the procedure will then fill a "Colonoscopy Report Form" including the number of polyps detected, size, shape, polypectomy method and cleanliness of the bowel.

The investigators did a pilot study with 150 subjects to check the mean no.of adenomas per colonoscopy, no.of adenomas detected in the right colon during the second look and to estimate the recruitment rate. Based on those results the investigators started this study with a large sample size. The investigators are planning to do an interim analysis after recruiting 450 subjects (30% of total enrollment). The results of the analysis will determine whether the investigators complete recruitment of the initially approved sample size of 1500 subjects.

ELIGIBILITY:
Inclusion Criteria:

* All increased risk patients (Patients with family history or personal history of colon polyps or colon cancer and FOBT positive) referred for a screening colonoscopy at the Forzani and MacPhail Colon Cancer Screening Centre will be considered for enrollment.

Exclusion Criteria:

* Average Risk patients
* Previous colon surgery
* Hereditary Polyposis Syndromes
* Suspected polyps or CRC before colonoscopy that have been suggested by another modality (Barium Enema, Virtual Colonoscopy, Flexible Sigmoidoscopy)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) in the right colon using High Definition White Light Colonoscopy Versus I-Scan enhanced Colonoscopy. | Colonoscopy report form provided to the Endoscopist will be filled out and collected after the procedure (1hour). All polyps reviewed by pathologist (1 week)
  Adenoma Detection Rate is defined as no. of colonoscopies at which one or more histologically confirmed adenomas were found divided by the total no. of colonoscopies performed in the same time period. The "Colonoscopy Report Form" filled by the Endoscopist helps to assess the number of polyps including an endoscopic description (Location, Size, Shape) of these lesions. Following formal review by the pathologist the polyp classification (eg: Whether it is an adenoma) is determined.

SECONDARY OUTCOMES:
Adenoma Detection Rate (ADR) in the right colon during the "Second Look" irrespective of imaging modality. | Second look in the right colon and finally withdrawing through the entire colon (approximately 5 min)
  The planned "Second Look" of the right colon will involve withdrawing from the cecum to hepatic flexure, then re-inserting to cecum and finally withdrawing through the entire colon. This is to determine if a "Second Look" in the right colon increases the ADR compared with a single inspection irrespective of imaging modality.
Adenoma Detection Rate (ADR) of High Definition White Light Colonoscopy Versus I-Scan colonoscopy through out the entire colon. | "Colonoscopy Report Form" provided to the endoscopist will be filled out and collected after the procedure (1 hour). All polyps reviewed by pathologist (1 week)
  Adenoma Detection Rate is defined as no. of colonoscopies at which one or more histologically confirmed adenomas were found divided by the total no. of colonoscopies performed in the same time period. The "Colonoscopy Report Form' completed by the Endoscopist helps to assess the number of polyps detected and an endoscopic description (location, shape, size) of these polyps.Following formal review by the pathologist the polyp classification (Eg: wether it is an Adenoma) is determined.

OTHER OUTCOMES:
Presence or absence of learning effect while using this technology | 12-18 months
  To determine if there is a learning effect when using this technology given that use of I-Scan may train the human eye to better identify adenomas even without image enhancement.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Robert Hilsden, MD, Principal Investigator — Faculty of Medicine, University of Calgary
Locations (1):
- Forzani & MacPhail Colon Cancer Screening Centre, Alberta Health Services, Calgary, Alberta, Canada